CLINICAL TRIAL: NCT04887831
Title: A Phase 2, Randomized, Open-Label Study of Trilaciclib Administered With First-Line Platinum-Based Chemotherapy and Avelumab Maintenance Therapy in Patients With Untreated, Locally Advanced or Metastatic Urothelial Carcinoma (PRESERVE 3)
Brief Title: Trilaciclib, a CDK 4/6 Inhibitor, in Patients With Advanced/Metastatic Bladder Cancer Receiving Chemotherapy Then Avelumab
Acronym: PRESERVE3
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor no longer pursuing trilaciclib for the indication.
Sponsor: G1 Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G1T28-209; 2021-000205-24 (EudraCT Number); IND: 156967 (Other: USFDA)
Record Dates: First submitted 2021-05-05; First posted 2021-05-14 (Actual); Results first posted 2025-08-17 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Urothelial Carcinoma; Bladder Cancer; Myelosuppression Adult; Chemotherapy-induced Neutropenia; Metastatic Bladder Cancer
Keywords: Trilaciclib dihydrochloride/Cosela; Metastatic Urothelial Carcinoma; Cyclin-dependent kinase 4/6 inhibitor; Immuno-oncology; Solid tumor; Chemotherapy-induced myelosuppression; Myeloprotective
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — trilaciclib; Gemcitabine; Cisplatin; Carboplatin; avelumab

STUDY DESIGN:
Intervention Model Description: Random assignment (1:1) to one of two treatment arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Platinum-based chemotherapy followed by avelumab maintenance therapy (Active Comparator): Gemcitabine 1000 milligram per square meter (mg/m^2) + Cisplatin (70 mg/m^2) or Carboplatin (Area under the concentration-time curve [AUC] 4.5) followed by Avelumab (800 mg)
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Drug: Carboplatin; Drug: Avelumab
- Trilaciclib plus platinum-based chemotherapy followed by avelumab maintenance therapy (Experimental): Trilaciclib (240 mg/m^2) + Gemcitabine (1000 mg/m^2) + Cisplatin (70 mg/m^2) or Carboplatin (AUC 4.5) followed by Trilaciclib (240 mg/m^2) + Avelumab (800 mg)
  Interventions: Drug: Trilaciclib; Drug: Gemcitabine; Drug: Cisplatin; Drug: Carboplatin; Drug: Avelumab

INTERVENTIONS:
Drug: Trilaciclib — Trilaciclib administered IV prior to chemotherapy and avelumab maintenance therapy on each day chemotherapy and avelumab maintenance therapy is administered.
  Other Names: Cosela; G1T28
  Arms: Trilaciclib plus platinum-based chemotherapy followed by avelumab maintenance therapy
Drug: Gemcitabine — Gemcitabine administered IV on Day 1 and Day 8 of each 21-day cycle
Drug: Cisplatin — Cisplatin administered IV on Day 1 of each 21-day cycle
Drug: Carboplatin — Carboplatin administered IV on Day 1 of each 21-day cycle
Drug: Avelumab — Avelumab administered IV on Day 1 of each 14-day maintenance cycle
  Other Names: Bavencio

SUMMARY:
This is a Phase 2, multicenter, randomized, open-label study evaluating the safety and efficacy of trilaciclib administered with platinum-based chemotherapy followed by trilaciclib administered with avelumab maintenance therapy compared with platinum-based chemotherapy followed by avelumab maintenance therapy in participants receiving first-line treatment for advanced/metastatic urothelial carcinoma.

DETAILED DESCRIPTION:
Participants will be randomly assigned (1:1) to receive standard of care platinum-based chemotherapy (with or without the addition of trilaciclib) administered intravenously (IV) in 21-day cycles followed by standard of care avelumab maintenance therapy (with or without the addition of trilaciclib) administered IV in 14-day cycles.

Participants enrolled in the study will be eligible to receive 4-6 cycles of platinum-based chemotherapy, and participants without progressive disease (PD) as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 guidelines (i.e., with an ongoing complete response [CR], partial response [PR], or stable disease [SD]) after platinum-based chemotherapy will be eligible to receive avelumab maintenance therapy until disease progression, unacceptable toxicity, withdrawal of consent, Investigator decision, or the end of the trial, whichever comes first.

Participants will be followed for survival approximately every 3 months after receiving the last dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Histologically documented, locally advanced (T4b, any N; or any T, N 2-3) or metastatic urothelial carcinoma (M1, Stage IV) (also termed Transitional cell carcinoma [TCC] or Urothelial cell carcinoma [UCC] of the urinary tract; including renal pelvis, ureters, urinary bladder, and urethra)

   1. Participants with mixed histologies are required to have a dominant transitional cell pattern (small cell carcinoma of any proportion is not allowed)
   2. Locally advanced bladder cancer must be inoperable on the basis of involvement of pelvic sidewall or adjacent viscera (clinical Stage T4b) or bulky nodal metastasis (N2-N3)
3. Measurable disease as defined by RECIST v1.1

   a. Previously irradiated lesions should not be counted as target lesions unless there has been demonstrated progression in the lesion since radiotherapy and no other lesions are available for selection as target lesions.
4. Considered to be eligible to receive platinum-based chemotherapy and avelumab maintenance therapy, in the Investigator's judgment
5. No prior systemic therapy in the inoperable, locally advanced, or metastatic setting including chemotherapy, immune checkpoint inhibitor therapy, targeted therapy, or investigational agents

   1. For participants who received prior adjuvant/neoadjuvant chemotherapy for urothelial carcinoma, a treatment-free interval > 12 months between the last treatment administration and the date of recurrence is required in order to be considered treatment-naïve in the metastatic setting. If a participant received adjuvant/neoadjuvant chemoradiation for urothelial carcinoma, a treatment-free interval >12 months between last platinum dose and the date of recurrence is required.
   2. For participants who received prior Immune checkpoint inhibitors (ICI) therapy in the adjuvant/neoadjuvant setting, a treatment-free interval > 3 months between the last dose of ICI and date of recurrence is required.
   3. Prior local intravesical chemotherapy or immunotherapy is allowed if completed ≥4 weeks prior to the initiation of study treatment
6. A formalin-fixed paraffin-embedded (FFPE) tumor tissue block (75-micron) or at least 15 (5-micron) unstained slides from archival or fresh tumor biopsy or resection; the most recent biopsy tissue preferred. Participants who have fewer than 15 unstained slides available at baseline (but no fewer than 10) may be eligible following discussion with the Medical Monitor.

   1. Tumor tissue should be of good quality based on total and viable tumor content. For core-needle biopsy specimens, at least three cores should be submitted for evaluation.
   2. Transurethral resection of bladder tumor (TURBT) specimens must contain a muscle -invasive component (i.e., T2 or greater) of the bladder tumor as verified by local pathology review. If the TURBT specimens do not contain a muscle-invasive component, then specimens obtained at the time of cystectomy/nephroureterectomy (i.e., pT2 or greater) or metastatic spread (i.e., a sample from a metastatic lesion) will be required prior to randomization. An archival specimen, if available, should also be submitted.
   3. Participants who do not have tissue specimens that meet eligibility requirements may undergo a biopsy during the screening period. Acceptable samples include core needle biopsies for deep tumor tissue (minimum three cores) or excisional, incisional, punch, or forceps biopsies for cutaneous, subcutaneous, or mucosal lesions.
   4. Tumor tissue from bone metastases is not evaluable for programmed death-ligand 1 (PD-L1) expression and is therefore not acceptable.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
8. Adequate organ function as demonstrated by the following laboratory values:

   1. Hemoglobin ≥9.0 gram per deciliter (g/dL) in the absence of RBC transfusion or ESA administration within 14 days prior to first dose of study drug
   2. Absolute neutrophil count (ANC) ≥1.5 × 10^9/L
   3. Platelet count ≥100 × 10^9/L
   4. Estimated glomerular filtration rate ≥ 30 mL/minute/1.73 m^2
   5. Total bilirubin ≤1.5 × upper limit of normal (ULN) (<3 ULN if Gilbert's disease)
   6. ALT and AST ≤2.5 × ULN in the absence of liver metastasis or <5 × ULN in the presence of liver metastasis
9. Resolution of nonhematologic toxicities from prior systemic therapy, radiation therapy, or surgical procedures to ≤ Grade 1

   a. Alopecia and sensory neuropathy ≤ Grade 2, as well as any electrolyte laboratory abnormalities not constituting a safety risk based on investigator's judgment are acceptable
10. Predicted life expectancy of ≥3 months
11. Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
12. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form and in this protocol

Exclusion Criteria:

1. Prior treatment with IL-2, IFN-α, anti-PD-L2, anti-CD137 or CD137 agonists, or cytotoxic T-lymphocyte associated protein 4 (CTLA-4) antibody (including ipilimumab), or any other therapeutic antibody or drug specifically targeting T cell co-stimulation or immune checkpoint pathways in any setting within 12 months prior to randomization
2. Malignancies other than urothelial carcinoma within 2 years prior to randomization, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ, or low-grade (Gleason ≤6) prostate cancer on surveillance without any plans for treatment intervention (e.g., surgery, radiation, or castration), or other non-clinically significant cancers, which may be considered after discussion with the medical monitor
3. Presence of central nervous system (CNS) metastases/leptomeningeal disease requiring immediate treatment with radiation therapy or steroids. Participant must be off steroids administered for brain metastases for at least 2 weeks prior to the first dose of study drugs. No stereotactic radiation within 1 week or whole-brain radiation within 14 days prior to first dose of study drugs
4. Uncontrolled ischemic heart disease or uncontrolled symptomatic congestive heart failure (≥ Class II New York Heart Association functional classification system), myocardial infarction within 6 months prior to first dose of study drugs, unstable angina, or serious cardiac arrhythmia requiring medication
5. QTcF interval > 480 msec. For participants with ventricular pacemakers, QTcF > 500 msec
6. Known history of stroke or cerebrovascular accident within 6 months prior to first dose of study drugs
7. Known history of serious, chronic active infection (e.g., human immunodeficiency virus, hepatitis B or C, tuberculosis, etc.)

   a. Viral load indicative of HIV, HIV 1/2 antibodies, positive hepatitis B virus surface antigen or hepatitis C virus ribonucleic acid (RNA) if anti-hepatitis C virus antibody screening test positive
8. Severe infections within 4 weeks prior to randomization, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia

   1. Therapeutic oral or IV antibiotic use within 2 weeks prior to randomization
   2. Participants receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease or for dental extraction) are eligible
9. Other uncontrolled serious chronic disease or psychiatric condition that in the Investigator's opinion could affect participant safety, compliance, or follow-up in the protocol
10. Receipt of any investigational medication within 4 weeks, or at least 5 half-lives, whichever is greater, prior to the first dose of study drugs
11. Known hypersensitivity or allergy to study drugs or any component in their formulations
12. Known severe hypersensitivity reactions to monoclonal antibodies (Grade ≥3), any history of anaphylaxis, or uncontrolled asthma (i.e., 3 or more features of asthma symptom control per Global Initiative for Asthma [GINA] 2020)
13. Prior hematopoietic stem cell or bone marrow transplantation, or solid organ transplantation
14. Radiotherapy to any non-Central nervous system (CNS) site within 1 week prior to the first dose of study drugs, or within 2 weeks to any CNS sites
15. Pregnant or lactating women

    a. Women of childbearing potential must have negative serum pregnancy test result within 7 days prior to initiating study treatment
16. Major surgical procedure, open biopsy, or significant traumatic injury within 4 weeks prior to study treatment start, or anticipation of the need for major surgical procedure during the course of the study
17. Received a live, attenuated vaccine within 4 weeks prior to the first dose of study drugs

    1. Inactive vaccines, including but not limited to influenza vaccine, pneumococcal vaccine, shingles vaccine, and regionally approved Covid-19 vaccines are allowed
    2. Participants must agree not to receive a live, attenuated influenza vaccine during study treatment
18. History of immune colitis, inflammatory bowel disease, idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest computed tomography (CT) scan

    a. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
19. Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent. Participants with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible
20. Current use of immunosuppressive medication, EXCEPT for the following:

    1. Intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection)
    2. Systemic corticosteroids at physiological doses ≤10 mg/day of prednisone or equivalent
    3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
21. Participants who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the Investigator, or participants who are employees of G1 Therapeutics, Inc. directly involved in the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2023-04-07 (Actual); Study Completion 2024-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical study director, Study Director — G1 Therapeutics, Inc.
Locations (34):
- United States (13):
  - Valkyrie Clinical Trial, Los Angeles, California
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - Rocky Mountain Cancer Centers, Littleton, Colorado
  - Florida Cancer Specialists - South, Fort Myers, Florida
  - Woodlands Medical Specialists, Pensacola, Florida
  - Florida Cancer Specialists - North, St. Petersburg, Florida
  - Beacon Cancer Center PLLC, Coeur d'Alene, Idaho
  - The Harry and Jeanette Weinberg Cancer Institute, Baltimore, Maryland
  - New York Oncology Hematology, P.C., Albany, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Northwest Cancer Specialists, P.C., Tigard, Oregon
  - Tennessee Oncology, PLLC, Nashville, Tennessee
- France (5):
  - Hopitaux Universitaires de Strasbourg - Service Oncologie et Hématologie, Strasbourg, Bas-Rhin
  - Institut Bergonié - Oncologie Médicale et Pédiatrique, Bordeaux, Gironde
  - Centre Léon Bérard - Département d'oncologie médicale, Lyon
  - Hôpital Européen Georges Pompidou - Service d'Oncologie Médicale, Paris
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
- Georgia (3):
  - High Technology Hospital MedCenter LTD, Batumi, Adjara
  - National Center of Urology Named after Laur Managadze, Tbilisi
  - LTD "Multiprofile Clinic Consilium Medulla", Tbilisi
- Hungary (3):
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz - Rendeloint, Szolnok, Jász-Nagykun-Szolnok
  - Országos Onkológiai Intézet, Budapest
  - Uzsoki Utcai Kórház, Budapest
- Spain (10):
  - Institut Català d'Oncologia-Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - ALTHAIA, Xarxa Assistencial Universitiria de Manresa, Manresa, Barcelona
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Vall d´Hebron, Barcelona
  - Hospital Clinic de Barcelona - Servicio de Oncología Médica, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - H.U. V. de las Nieves, Granada
  - Hospital Universitario Lucus Augusti, Lugo
  - Fundación Instituto Valenciano de Oncología, Valencia
  - Hospital Politecnic Universitari La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 55 sites in the United States (US), Hungary, Georgia, France, and Spain from 4 June 2021 (first participant enrolled) to 1 March 2024 (last participant last visit).
Pre-assignment Details: Of the 116 participants enrolled, 24 were screen failures and 92 participants were randomized to treatment.
Groups:
- Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy: Gemcitabine (1000 mg/m^2) + Cisplatin (70 mg/m^2) or Carboplatin (AUC 4.5) followed by Avelumab (800 mg)
  Gemcitabine: Gemcitabine administered IV on Day 1 and Day 8 of each 21-day cycle
  Cisplatin: Cisplatin administered IV on Day 1 of each 21-day cycle
  Carboplatin: Carboplatin administered IV on Day 1 of each 21-day cycle
  Avelumab: Avelumab administered IV on Day 1 of each 14-day maintenance cycle
Period: Overall Study
Arm/Group | Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy | Trilaciclib Plus Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy
Started | 47 | 45
Completed | 0 | 0
Not Completed | 47 | 45
Not completed — Death | 26 | 26
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Study Terminated by Sponsor | 18 | 17
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy | Trilaciclib Plus Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy | Total
Number analyzed (Participants) | 47 | 45 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 17 | 30
  >=65 years | 34 | 28 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (10.34) | 67.3 (8.40) | 67.6 (9.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 39 | 34 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 38 | 34 | 72
  Unknown or Not Reported | 8 | 9 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 37 | 34 | 71
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 11 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression-Free Survival (PFS) During Overall Study
Description: The PFS was defined as the time from date of randomization to the date of the first documented disease progression, or death in the absence of PD for those who had a PFS event, and the time from randomization to the censoring date for those who did not have a PFS event.
Time Frame: From date of randomization until date of documented radiologic disease progression per RECIST v1.1 or death due to any cause, whichever comes first. Approximately 96 weeks
Population: The Intent-to-treat (ITT) analysis set included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy | Trilaciclib Plus Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy
Number analyzed (Participants) | 47 | 45
Participants | 36 | 34

2. Secondary Outcome: Number of Participants With Objective Response Rate (ORR) During Chemotherapy Period
Description: The ORR defined as the percentage of participants who had an objective response (unconfirmed or confirmed) per RECIST v1.1
Time Frame: as for outcome 1
Population: The Response Evaluable (RE) analysis set included those participants who were in the ITT population and received at least 1 dose of any study drug, have measurable (target) tumor lesion(s) at baseline tumor assessment, and have at least 1 of the following: (1) at least 1 post-baseline tumor assessment; (2) discontinued treatment because of clinical progression prior to their first post-baseline tumor scan; (3) died due to disease progression prior to their first post-baseline tumor scan.
Measure: Count of Participants; unit: Participants
Arm/Group | Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy | Trilaciclib Plus Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy
Number analyzed (Participants) | 46 | 45
Participants | 24 | 19
Statistical Analysis 1: Comparison: Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy vs Trilaciclib Plus Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy; Test type: Other; p = 0.340, Cochran-Mantel-Haenszel — The 2-sided p-value was calculated using stratified CMH method to account for the presence of visceral metastasis (yes/no) and initial chemotherapy type (cisplatin/carboplatin) as the stratification factors; Adjusted percentage difference = -0.101, 95% CI 2-sided [-0.308 to 0.105], Standard Error of Mean 0.1052

3. Secondary Outcome: Number of Participants With Objective Response Rate During Overall Treatment Period
Description: as for outcome 2
Time Frame: as for outcome 1
Population: The RE analysis set included those participants who were in the ITT population and received at least 1 dose of any study drug, have measurable (target) tumor lesion(s) at baseline tumor assessment, and have at least 1 of the following: (1) at least 1 post-baseline tumor assessment; (2) discontinued treatment because of clinical progression prior to their first post-baseline tumor scan; (3) died due to disease progression prior to their first post-baseline tumor scan.
Measure: Count of Participants; unit: Participants
Arm/Group | Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy | Trilaciclib Plus Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy
Number analyzed (Participants) | 46 | 45
Participants | 24 | 23
Statistical Analysis 1: Comparison: Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy vs Trilaciclib Plus Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy; Test type: Other; p = 0.938, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Adjusted percentage difference = -0.008, 95% CI 2-sided [-0.220 to 0.203], Standard Error of Mean 0.1078

4. Secondary Outcome: Percentage of Participants Survived at 12 Months [Overall Survival (OS) Rate]
Description: The OS during the study was defined as the time from the date of randomization to the date of death for participants who died in the study regardless of cause, or to the last contact date known to be alive for those who survived as of the date of data snapshot for intermediate planned analysis or final database lock for final analyses (censored cases).
Time Frame: From date of randomization (Day 1) up to Month 12
Population: The ITT analysis set included all randomized participants.
Measure: Number; unit: Percentage Of - Participants
Arm/Group | Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy | Trilaciclib Plus Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy
Number analyzed (Participants) | 47 | 45
Percentage Of - Participants | 64.6 | 54.0

5. Secondary Outcome: Myeloprotective Effects
Description: To assess the effects of trilaciclib on the neutrophil lineage as measured by the occurrence of severe neutropenia during platinum-based chemotherapy treatment. Myeloprotective effects protect the blood-forming cells in the bone marrow from the side effects of chemotherapy such as bone marrow suppression.
Time Frame: Cycle 1 Day 1 (each cycle is 21 days) through treatment with platinum-based chemotherapy, approximately up to 4 months
Population: The ITT analysis set included all randomized participants.
Measure: Mean (Standard Deviation); unit: Duration of severe neutropenia (days)
Arm/Group | Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy | Trilaciclib Plus Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy
Number analyzed (Participants) | 47 | 45
Duration of severe neutropenia (days) | 0.8 (2.88) | 0.5 (2.00)

6. Secondary Outcome: Disease Control Rate (DCR) During Maintenance Period
Description: The DCR was defined as the percentage of participants with best overall response (BOR) of confirmed CR, confirmed PR, or SD.
Time Frame: From date of randomization, up to 12 cycles (21-day each) of Maintenance therapy until disease progression, unacceptable toxicity or discontinuation by the participant or investigator, assessed up to 34 weeks.
Population: The maintenance population included all the randomized participants who received at least 1 dose of any study drug during the maintenance period.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy | Trilaciclib Plus Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy
Number analyzed (Participants) | 29 | 30
Percentage of participants | 44.8 [26.4 to 64.3] | 26.7 [12.3 to 45.9]

7. Secondary Outcome: Disease Control Rate During Overall Study
Description: The DCR was defined as the percentage of participants with BOR of confirmed CR, confirmed PR, or SD.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy | Trilaciclib Plus Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy
Number analyzed (Participants) | 46 | 45
percentage of participants | 89.1 [76.4 to 96.4] | 82.2 [67.9 to 92.0]

8. Secondary Outcome: Duration of Response (DoR), Overall Study
Description: The DoR was defined as the time from the date of first documented response (CR or PR) to date of first occurrence of disease progression as determined by the investigator, or death from any cause, whichever occurs first.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy | Trilaciclib Plus Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy
Number analyzed (Participants) | 46 | 45
Months | 6.6 [3.3 to 8.3] | 7.0 [4.7 to 15.6]

9. Secondary Outcome: Number of Participants With Progression-Free Survival During Maintenance Period
Description: as for outcome 1
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy | Trilaciclib Plus Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy
Number analyzed (Participants) | 29 | 30
Participants | 22 | 20

10. Secondary Outcome: Percentage of Participants With Probability of Survival at 16 Months.
Description: The OS was defined as the time from the date of randomization to the date of death for participants who died in the study regardless of cause, or to the last contact date known to be alive for those who survived as of the date for final database lock (censored cases).
Time Frame: 16 months
Population: The ITT analysis set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy | Trilaciclib Plus Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy
Number analyzed (Participants) | 47 | 45
percentage of participants | 44.5 [29.8 to 58.2] | 46.9 [31.5 to 60.8]

11. Secondary Outcome: Overall Survival During Maintenance Period
Description: The OS was calculated as the time (months) from date of randomization to the date of death due to any cause.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy | Trilaciclib Plus Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy
Number analyzed (Participants) | 29 | 30
Participants | 13 | 17

12. Secondary Outcome: Overall Survival During Overall Study
Description: The OS was calculated as the time (months) from date of randomization to the date of death due to any cause.
Time Frame: From first administration of study treatment (Day 1) until 30 days after the last dose of study treatment, approximately 96 weeks.
Population: The ITT analysis set included all randomized participants.
Measure: Median (Full Range); unit: months
Arm/Group | Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy | Trilaciclib Plus Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy
Number analyzed (Participants) | 47 | 45
months | 14.6 [10.5 to NA] — CI upper limit for the median OS could not be estimated due to an insufficient number of patients with events as a result of insufficient follow-up time and censoring due to early study termination. | 15.4 [10.2 to NA] — CI upper limit for the median OS could not be estimated due to an insufficient number of patients with events as a result of insufficient follow-up time and censoring due to early study termination.

13. Secondary Outcome: Number of Participants With Adverse Events (AE)
Description: An AE was defined as any untoward or unfavourable medical occurrence in a clinical research study participant, including any abnormal sign (e.g. abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participants' involvement in the research, whether or not considered related to participation in the research.
Time Frame: as for outcome 12
Population: The Safety Population included all randomized participants who received at least 1 dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy | Trilaciclib Plus Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy
Number analyzed (Participants) | 47 | 45
Participants | 45 | 44

14. Secondary Outcome: Number of Participants With Serious Adverse Events (SAE)
Description: SAEs were defined as any untoward medical occurrence that at any dose resulted in death, was life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity or was a congenital anomaly/birth defect.
Time Frame: as for outcome 12
Population: The Safety Population included all randomized participants who received at least 1 dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy | Trilaciclib Plus Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy
Number analyzed (Participants) | 47 | 45
Participants | 13 | 18

ADVERSE EVENTS:
Time Frame: From first administration of study treatment (Day 1) until 30 days after the last dose of study treatment, approximately 96 weeks.
Description: The Safety Population included all randomized participants who received at least 1 dose of any study drug.
Arm/Group | Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy | Trilaciclib Plus Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy
All-Cause Mortality (participants affected / at risk) | 26/47 | 26/45
Serious Adverse Events (participants affected / at risk) | 13/47 | 18/45
Other Adverse Events (participants affected / at risk) | 45/47 | 44/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy (N=47) | Trilaciclib Plus Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy (N=45)
Optic Neuritis (Nervous system disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Immue-mediated adverse reaction (Immune system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 3
Haematuria (Renal and urinary disorders) | 2 | 1
Asthenia (General disorders) | 1 | 1
Sepsis (Infections and infestations) | 1 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Septic Shock (Infections and infestations) | 1 | 3
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 3
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Muscle necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 2
Urosepsis (Infections and infestations) | 1 | 2
Cerebral thrombosis (Nervous system disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Klebsiella infection (Infections and infestations) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy (N=47) | Trilaciclib Plus Platinum-based Chemotherapy Followed by Avelumab Maintenance Therapy (N=45)
Anaemia (Blood and lymphatic system disorders) | 28 | 25
Neutropenia (Blood and lymphatic system disorders) | 16 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 10 | 8
Leukopenia (Blood and lymphatic system disorders) | 5 | 1
Asthenia (General disorders) | 13 | 13
Fatigue (General disorders) | 10 | 10
Pyrexia (General disorders) | 5 | 6
Oedema peripheral (General disorders) | 5 | 2
Pain (General disorders) | 2 | 4
Mucosal inflammation (General disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 18 | 22
Constipation (Gastrointestinal disorders) | 13 | 7
Diarrhoea (Gastrointestinal disorders) | 6 | 5
Vomiting (Gastrointestinal disorders) | 4 | 7
Abdominal pain upper (Gastrointestinal disorders) | 0 | 6
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Dry mouth (Gastrointestinal disorders) | 3 | 1
Platelet count decreased (Investigations) | 10 | 4
Neutrophil count decreased (Investigations) | 9 | 4
Blood creatinine increased (Investigations) | 3 | 5
Blood alkaline phosphatase increased (Investigations) | 3 | 2
Weight decreased (Investigations) | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 9 | 14
Hypomagnesaemia (Metabolism and nutrition disorders) | 9 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 0
COVID-19 (Infections and infestations) | 4 | 6
Urinary tract infection (Infections and infestations) | 4 | 6
Respiratory tract infection (Infections and infestations) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Dysgeusia (Nervous system disorders) | 7 | 2
Headache (Nervous system disorders) | 4 | 3
Neuropathy peripheral (Nervous system disorders) | 2 | 4
Dizziness (Nervous system disorders) | 1 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3
Insomnia (Psychiatric disorders) | 6 | 5
Tinnitus (Ear and labyrinth disorders) | 4 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Haematuria (Renal and urinary disorders) | 5 | 5
Renal failure (Renal and urinary disorders) | 0 | 6
Renal impairment (Renal and urinary disorders) | 0 | 3

LIMITATIONS AND CAVEATS:
This study was terminated earlier than initially proposed by the Sponsor for non-safety related reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator agrees to submit any disclosure to Sponsor for review at least thirty (30) days prior to submission. Within sixty (60) days of its receipt, Sponsor can provide feedback on any disclosure Sponsor may require Investigator to remove, Confidential Information (other than study data), and/or to delay the proposed publication or presentation for an additional sixty (60) days to enable Sponsor to seek patent protection for inventions.

DOCUMENTS (2):
  • Study Protocol (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/31/NCT04887831/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-06): https://cdn.clinicaltrials.gov/large-docs/31/NCT04887831/SAP_001.pdf